CLINICAL TRIAL: NCT04213027
Title: Sacrospinous Ligament Fixation vs. Ischial Spine Fasicia Fixation With Conventional Surgical Instruments in Chinese Apical Prolapse Female Patients: a Multi-center, Prospective, Randomized Clinical Trial
Brief Title: RCT for SSLF vs. ISFF With Conventional Surgical Instruments in Chinese Apical Prolapse Female Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, zhulan, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUMCH SSLFvsISFF-CSI
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Apical Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSLF-CSI (Active Comparator): native tissue repair procedure with conventional surgical instruments in Chinese apical prolapse female patients randomized to Sacrospinous ligament fixation (SSLF) .
  Interventions: Procedure: native tissue repair procedures with conventional surgical instruments
- ISFF-CSI (Active Comparator): native tissue repair procedure with conventional surgical instruments in Chinese apical prolapse female patients randomized to Ischial spinous fascia fixation (ISFF)
  Interventions: Procedure: native tissue repair procedures with conventional surgical instruments

INTERVENTIONS:
Procedure: native tissue repair procedures with conventional surgical instruments — Sacrospinous ligament fixation (SSLF): treatment for apical prolapse with vaginal fornix suspended to sacrospinous ligament; Ischial spinous fascia fixation (ISFF): treatment for apical prolapse with vaginal fornix suspended to ischial spinous fascia (ISFF).

SUMMARY:
This trial is designed to investigate the efficacy and safety of two native tissue repair procedure with conventional surgical instruments in Chinese apical prolapse female patients (POP-Q II-IV) and compare the outcome in prolapse women randomized to Sacrospinous ligament fixation (SSLF) and Ischial spinous fascia fixation (ISFF).

DETAILED DESCRIPTION:
The population will include Chinese female patients with advanced apical prolapse (stage II-III) and who are undergoing Sacrospinous Ligament Fixation (SSLF) and Ischial spinous fascia fixation (ISFF) procedure using conventional surgical instruments without special instrument. After enrollment, standardized baseline data including demographics, POPQ evaluation, series of validated questionaires via interviews( PFDI-20, PFIQ-7, PISQ-12) will be collected by study personnel at the baseline visit. Eligible consenting patients will proceed to randomizations with equal probability of assignment to SSLF or ISFF. Randomization to either SSLF or ISFF will take place preoperatively by each clinical site using a random permutated block design. After index surgical intervention, scheduled follow-up will occur at 3, 6, 12, 24 and 36 months after the index surgery. At the follow-up visits, POPQ examination will be performed and an update of current medications, an assessment of new or continuing pelvic floor disorders, adverse events that occurred since the previous evaluation, and an assessment of health care costs. A series of validated instruments will be administered via interviews to including PFDI-20, PFIQ-7, PISQ-12, PGI-C.

ELIGIBILITY:
Inclusion Criteria:

1. Women with apical prolapse with POP-Q II-IV (but no anterior wall prolapse stage IV)
2. SSLF or ISFF is proceeded as described before，while ancillary procedures like vaginal hysterectomy, anterior/posterior vaginal wall repair without mesh or mid-urethral suspension could be performed simultaneously.
3. Women who have been eligible for long-term follow-up.
4. Women who agreed to participate in the study and signed informed consent.

Exclusion Criteria:

1. Women who have surgical history for prolapse with mesh.
2. Women who have contraindication for surgical procedure
3. Women who are unable to comply with the study procedures

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of surgical success | up to 36 months after operation
  definition for surgical success is symptomatic prolapse below grade II occurred at 3 months after operation, and the severest indication point in POP-Q evaluation was taken as the criterion. No vaginal swelling sensation, that is answer "no" for PFDI-20 Questionnaire Question 3, "Do you often see or feel vaginal tumors come out?".
  The patient's self-perception symptoms is improved or improved significantly, that is answer 1 or 2 for the PGI-C questionnaire.
  There is no need of further treatment for prolapse, such as reoperation or pessary.

SECONDARY OUTCOMES:
rate of Postoperative recurrence | from 3 months after operation up to 36 months after operation
  definition for postoperative recurrence is symptomatic prolapse above grade II occurred 3 months after operation, and the severest indication point in POP-Q evaluation was taken as the criterion. Vaginal swelling sensation, that is answer "yes" for PFDI-20 Questionnaire Question 3, "Do you often see or feel vaginal tumors come out?".
  There is need of further treatment for prolapse, such as reoperation or pessary.
visual analogue scales | up to 36 months after operation, usuallly within 3 days after operation
  postoperative pain evaluation esp. hip pain by visual analogue scales (VAS). Visual Analogue Scale (VAS) is a self-report measure consisting simply of a 10 centimeter line with a statement at each end representing one extreme of the dimension being measured (most often intensity of pain). VAS result will be reported ranging from 0 to 10, with 0 representing no pain, and 10 representing unbearable severe pain
changes between preoperative and postoperative symptomatic improvement using validated instruments(PFIQ-7) | up to 36 months after operation
  Relief of symptoms using validated instruments, pelvic floor impact questionnaire short form 7(PFIQ-7)。PFIQ-7 scores 0-300, the higher the severer negative influence on patient.
changes between preoperative and postoperative symptomatic improvement using validated instruments(PFDI-20) | up to 36 months after operation
  Relief of symptoms using validated instruments, pelvic floor distress inventory short form 20(PFDI-20), PFDI-20 scores 0-300, the higher the severer negative influence on patient.
changes between preoperative and postoperative symptomatic improvement using validated instruments(PISQ-12) | up to 36 months after operation
  Relief of symptoms using validated instruments, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form(PISQ-12), PISQ-12 scores 0-48, the higher, the severer negative influence on patient.
results of postoperative symptomatic improvement using patient global impression of change (PGI-C) | up to 36 months after operation
  Relief of symptoms using patient global impression of change (PGI-C)， PGI-C scores 1-7, the higher, the the severer negative influence on patient.
intraoperative and post operative complications | up to 36 months after operation
  using IUGA/ICS joint terminology CTS coding system and dingo system

CONTACTS AND LOCATIONS:
Overall Officials: Yongxian Lu, Principal Investigator — 1st Affiliated hospital of PLA general hospital; Zhiyuan Dai, Principal Investigator — Shanghai First Maternity and Infant Hospital; Wenyan Wang, Principal Investigator — 2nd Affiliated hospital of Anhui Medical college; Zhaoai Li, Principal Investigator — Shan'xi Province Women's and Children's Hospital; Yuling Wang, Principal Investigator — Foshan Women's and Children's Hospital; Shunyu Hou, Principal Investigator — Suzhou City Hospital; Xiangjuan Li, Principal Investigator — Hangzhou Women's and Children's Hospital; Lubin Liu, Principal Investigator — Chongqing Women's and Children's Hospital; Le Ma, Principal Investigator — Beijing Obstetrics and Gynecology Hospital; Tao Xu, Principal Investigator — Statistics Department of Peking Union Medical College; Joseph Schaffer, Principal Investigator — University of Texas Southwestern Medical Center; Marko J Jachtorowycz, Principal Investigator — Saint Francis Hospital; Lan Zhu, Study Chair — Peking Union Medical College Hospital; Yuxin Dai, Study Director — Peking Union Medical College Hospital
Locations (5):
- China (5):
  - 2nd Affiliated hospital of Anhui Medical college, Hefei, Anhui
  - 1st Affiliated hospital of PLA general hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Suzhou City Hospital, Suzhou, Jiangsu
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014. doi: 10.1002/14651858.CD004014.pub5. PMID 23633316
- [Background] Barber MD, Maher C. Apical prolapse. Int Urogynecol J. 2013 Nov;24(11):1815-33. doi: 10.1007/s00192-013-2172-1. PMID 24142057
- [Background] Zhu L, Lang J, Zhang Q. Clinical study of ischia spinous fascia fixation--a new pelvic reconstructive surgery. Int Urogynecol J. 2011 Apr;22(4):499-503. doi: 10.1007/s00192-010-1307-x. PMID 21060988
- [Background] Ren C, Song XC, Zhu L, Ai FF, Shi HH, Sun ZJ, Chen J, Lang JH. [Prospective cohort study on the outcomes of sacrospinous ligament fixation using conventional instruments in treating stage Ⅲ-Ⅳ pelvic organ prolapse]. Zhonghua Fu Chan Ke Za Zhi. 2017 Jun 25;52(6):369-373. doi: 10.3760/cma.j.issn.0529-567X.2017.06.003. Chinese. PMID 28647958
- [Result] Haya N, Baessler K, Christmann-Schmid C, de Tayrac R, Dietz V, Guldberg R, Mascarenhas T, Nussler E, Ballard E, Ankardal M, Boudemaghe T, Wu JM, Maher CF. Prolapse and continence surgery in countries of the Organization for Economic Cooperation and Development in 2012. Am J Obstet Gynecol. 2015 Jun;212(6):755.e1-755.e27. doi: 10.1016/j.ajog.2015.02.017. Epub 2015 Feb 25. PMID 25724403